CLINICAL TRIAL: NCT03438812
Title: The Role of Dehydroepiandrosterone in the Maintenance of Mitochondrial Quality of Cumulus Cells in Poor Ovarian Responders
Brief Title: Dehydroepiandrosterone Maintain Mitochondrial Quality of Cumulus Cells in Poor Ovarian Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Visiting Staff, Department of Obstetrics and Gynecology, Principal Investigator, Clinical Lecturer, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS14-CT10-16
Record Dates: First submitted 2018-02-04; First posted 2018-02-20 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Poor Responders; Dehydroepiandrosterone
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Poor ovarian responders with DHEA (Experimental): Women who meet the Bologna criteria receive dehydroepiandrosterone (DHEA, 90 mg daily for two months at least) supplementation prior to the IVF cycle.
  Interventions: Dietary Supplement: dehydroepiandrosterone (DHEA)
- Poor ovarian responders (No Intervention): Women who meet the Bologna criteria undergo the IVF cycle without pretreatment with DHEA
- Normal ovarian responders (No Intervention): Women who do not meet the Bologna criteria and have normal ovarian response to ovarian stimulation.

INTERVENTIONS:
Dietary Supplement: dehydroepiandrosterone (DHEA) — Participants take DHEA 90 mg daily for two months at least before in vitro fertilization cycles.
  Arms: Poor ovarian responders with DHEA

SUMMARY:
To investigate whether the DHEA supplementation could improve mitochondrial quality in poor ovarian responders

DETAILED DESCRIPTION:
Women who underwent in vitro fertilization (IVF) treatment participated, including normal ovarian responders (NORs) and poor ovarian responders (PORs). PORs were assigned to receive DHEA supplementation or not before the IVF cycle. For all patients, cumulus cells (CCs) were obtained after oocyte retrieval. In the CCs, mRNA expression of mitochondria-related genes was measured. To compare the mRNA expression of mitochondria-related genes in the CCs among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Poor ovarian responders met the Bologna criteria, having at least two of the three following features: (1) advanced maternal age (≥ 40 years) or any other risk factor for POR, (2) a previous POR (≤ 3 oocytes with a conventional stimulation protocol), and (3) an abnormal ovarian reserve test. An abnormal ovarian reserve test was defined as antral follicle counts (AFC) < 5 or anti-Müllerian hormone (AMH) < 1 ng/mL in this study.
* Normal ovarian responders met the following criteria: (1) AFCs ≥ 5 or AMH ≥ 1 ng/mL and (2) the number of retrieved oocytes was between 5 and 15.

Exclusion Criteria:

* previous oophorectomy
* exposure to cytotoxic or pelvic irradiation for malignancy
* positive screening for recurrent pregnancy loss (chromosome mapping, antinuclear antibodies, extractable nuclear antigens, antiphospholipid antibodies, thrombophilic screening)
* any other sensitizing or ovarian stimulating therapy during the previous 3 months

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
mitochondria related genes expression | through study completion, an average of 1 year
  cumulus cells genes expression

SECONDARY OUTCOMES:
oocytes | through study completion, an average of 1 year
  retrieved oocytes in number
embryos | numbers will be confirmed 3 days after fertilization
  day 3 embryos in number
pregnancy rate | pregnancy will be confirmed 4 weeks after embryo transfer
  clinical pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Ph.D., Study Director — Kaohsiung Veterans General Hospital.; Li-Te Lin, Ph.D., Principal Investigator — Kaohsiung Veterans General Hospital.; Salvatore Giovanni Vitale, M.D., Principal Investigator — University of Messina
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Lin LT, Tsui KH, Wang PH. Clinical application of dehydroepiandrosterone in reproduction: A review of the evidence. J Chin Med Assoc. 2015 Aug;78(8):446-53. doi: 10.1016/j.jcma.2014.12.008. Epub 2015 Feb 20. PMID 25708822
- [Background] Zhang J, Qiu X, Gui Y, Xu Y, Li D, Wang L. Dehydroepiandrosterone improves the ovarian reserve of women with diminished ovarian reserve and is a potential regulator of the immune response in the ovaries. Biosci Trends. 2015 Dec;9(6):350-9. doi: 10.5582/bst.2015.01154. PMID 26781792
- [Background] Nagels HE, Rishworth JR, Siristatidis CS, Kroon B. Androgens (dehydroepiandrosterone or testosterone) for women undergoing assisted reproduction. Cochrane Database Syst Rev. 2015 Nov 26;2015(11):CD009749. doi: 10.1002/14651858.CD009749.pub2. PMID 26608695
- [Background] Tsui KH, Lin LT, Horng HC, Chang R, Huang BS, Cheng JT, Wang PH. Gene expression of cumulus cells in women with poor ovarian response after dehydroepiandrosterone supplementation. Taiwan J Obstet Gynecol. 2014 Dec;53(4):559-65. doi: 10.1016/j.tjog.2014.09.003. PMID 25510701
- [Background] Lin LT, Wang PH, Chen SN, Li CJ, Wen ZH, Cheng JT, Tsui KH. Protection of cumulus cells following dehydroepiandrosterone supplementation. Gynecol Endocrinol. 2017 Feb;33(2):100-104. doi: 10.1080/09513590.2016.1214262. Epub 2016 Aug 12. PMID 27684542
- [Background] Santos TA, El Shourbagy S, St John JC. Mitochondrial content reflects oocyte variability and fertilization outcome. Fertil Steril. 2006 Mar;85(3):584-91. doi: 10.1016/j.fertnstert.2005.09.017. PMID 16500323
- [Background] Zeng HT, Ren Z, Yeung WS, Shu YM, Xu YW, Zhuang GL, Liang XY. Low mitochondrial DNA and ATP contents contribute to the absence of birefringent spindle imaged with PolScope in in vitro matured human oocytes. Hum Reprod. 2007 Jun;22(6):1681-6. doi: 10.1093/humrep/dem070. Epub 2007 Apr 20. PMID 17449512
- [Background] Lee SK, Zhao MH, Kwon JW, Li YH, Lin ZL, Jin YX, Kim NH, Cui XS. The association of mitochondrial potential and copy number with pig oocyte maturation and developmental potential. J Reprod Dev. 2014 Apr 24;60(2):128-35. doi: 10.1262/jrd.2013-098. Epub 2014 Feb 4. PMID 24492657
- [Background] Zhang M, Niu W, Wang Y, Xu J, Bao X, Wang L, Du L, Sun Y. Dehydroepiandrosterone treatment in women with poor ovarian response undergoing IVF or ICSI: a systematic review and meta-analysis. J Assist Reprod Genet. 2016 Aug;33(8):981-91. doi: 10.1007/s10815-016-0713-5. Epub 2016 Apr 19. PMID 27094195
- [Background] Alexaki VI, Charalampopoulos I, Panayotopoulou M, Kampa M, Gravanis A, Castanas E. Dehydroepiandrosterone protects human keratinocytes against apoptosis through membrane binding sites. Exp Cell Res. 2009 Aug 1;315(13):2275-83. doi: 10.1016/j.yexcr.2009.04.006. Epub 2009 Apr 18. PMID 19379733
- [Background] Liu D, Si H, Reynolds KA, Zhen W, Jia Z, Dillon JS. Dehydroepiandrosterone protects vascular endothelial cells against apoptosis through a Galphai protein-dependent activation of phosphatidylinositol 3-kinase/Akt and regulation of antiapoptotic Bcl-2 expression. Endocrinology. 2007 Jul;148(7):3068-76. doi: 10.1210/en.2006-1378. Epub 2007 Mar 29. PMID 17395704
- [Background] Charalampopoulos I, Tsatsanis C, Dermitzaki E, Alexaki VI, Castanas E, Margioris AN, Gravanis A. Dehydroepiandrosterone and allopregnanolone protect sympathoadrenal medulla cells against apoptosis via antiapoptotic Bcl-2 proteins. Proc Natl Acad Sci U S A. 2004 May 25;101(21):8209-14. doi: 10.1073/pnas.0306631101. Epub 2004 May 17. PMID 15148390
- [Background] Ding X, Wang D, Li L, Ma H. Dehydroepiandrosterone ameliorates H2O2-induced Leydig cells oxidation damage and apoptosis through inhibition of ROS production and activation of PI3K/Akt pathways. Int J Biochem Cell Biol. 2016 Jan;70:126-39. doi: 10.1016/j.biocel.2015.11.018. Epub 2015 Nov 28. PMID 26643608
- [Background] Patel MA, Katyare SS. Effect of dehydroepiandrosterone (DHEA) treatment on oxidative energy metabolism in rat liver and brain mitochondria. A dose-response study. Clin Biochem. 2007 Jan;40(1-2):57-65. doi: 10.1016/j.clinbiochem.2006.08.014. Epub 2006 Sep 14. PMID 17052700
- [Background] Patel MA, Katyare SS. Treatment with dehydroepiandrosterone (DHEA) stimulates oxidative energy metabolism in the cerebral mitochondria. A comparative study of effects in old and young adult rats. Neurosci Lett. 2006 Jul 10;402(1-2):131-6. doi: 10.1016/j.neulet.2006.03.057. Epub 2006 Apr 19. PMID 16630690
- [Background] Boucret L, Chao de la Barca JM, Moriniere C, Desquiret V, Ferre-L'Hotellier V, Descamps P, Marcaillou C, Reynier P, Procaccio V, May-Panloup P. Relationship between diminished ovarian reserve and mitochondrial biogenesis in cumulus cells. Hum Reprod. 2015 Jul;30(7):1653-64. doi: 10.1093/humrep/dev114. Epub 2015 May 20. PMID 25994667
- [Background] Ogino M, Tsubamoto H, Sakata K, Oohama N, Hayakawa H, Kojima T, Shigeta M, Shibahara H. Mitochondrial DNA copy number in cumulus cells is a strong predictor of obtaining good-quality embryos after IVF. J Assist Reprod Genet. 2016 Mar;33(3):367-371. doi: 10.1007/s10815-015-0621-0. Epub 2016 Jan 9. PMID 26749386
- [Background] Tsai HD, Hsieh YY, Hsieh JN, Chang CC, Yang CY, Yang JG, Cheng WL, Tsai FJ, Liu CS. Mitochondria DNA deletion and copy numbers of cumulus cells associated with in vitro fertilization outcomes. J Reprod Med. 2010 Nov-Dec;55(11-12):491-7. PMID 21291035
- [Background] Au HK, Yeh TS, Kao SH, Tzeng CR, Hsieh RH. Abnormal mitochondrial structure in human unfertilized oocytes and arrested embryos. Ann N Y Acad Sci. 2005 May;1042:177-85. doi: 10.1196/annals.1338.020. PMID 15965061